CLINICAL TRIAL: NCT00003587
Title: Randomized Phase II Trial of Carboplatin/Gemcitabine Followed By Paclitaxel or Cisplatin/Vinorelbine Followed by Docetaxel in Advanced Non-Small Cell Lung Cancer
Brief Title: S9806: Combination Chemotherapy in Treating Patients With Stage IIIB or Stage IV Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066656; S9806 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 1999-11-01; First posted 2004-09-13 (Estimated); Last update posted 2012-10-08 (Estimated); Status verified 2012-10

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; squamous cell lung cancer; large cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; adenocarcinoma of the lung
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung | interventions — Carboplatin; Cisplatin; Docetaxel; Gemcitabine; Paclitaxel; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- carboplatin/gemcitabine/paclitaxel (Experimental): IV carboplatin AUC=5.5 day 1 every 21 days X 3 IV gemcitabine 1,000 mg/m^2/day, days 1 and 8 every 21 days X3 IV paclitaxel 225 mg/m^2/day, day 1 every 21 days X 3
  Interventions: Drug: carboplatin; Drug: gemcitabine; Drug: paclitaxel
- cisplatin/vinorelbine/docetaxel (Experimental): IV cisplatin 100 mg/m^2 day 1 every 21 days X 3 IV vinorelbine 25 mg/m^2/day, days 1 and 8 every 21 days X 3 IV docetaxel 75 mg/m^2 day 1 every 21 days X 3
  Interventions: Drug: cisplatin; Drug: docetaxel; Drug: vinorelbine

INTERVENTIONS:
Drug: carboplatin — AUC=5.5 day 1 every 21 days X 3
  Other Names: carbo
  Arms: carboplatin/gemcitabine/paclitaxel
Drug: cisplatin — IV cisplatin 100 mg/m^2 day 1 every 21 days X 3
  Other Names: platinol
  Arms: cisplatin/vinorelbine/docetaxel
Drug: docetaxel — IV docetaxel 75 mg/m^2 day 1 every 21 days X 3
  Other Names: taxotere
  Arms: cisplatin/vinorelbine/docetaxel
Drug: gemcitabine — IV gemcitabine 1,000 mg/m^2/day, days 1 and 8 every 21 days X3
  Other Names: gemzar
  Arms: carboplatin/gemcitabine/paclitaxel
Drug: paclitaxel — IV paclitaxel 225 mg/m^2/day, day 1 every 21 days X 3
  Other Names: taxol
  Arms: carboplatin/gemcitabine/paclitaxel
Drug: vinorelbine — IV vinorelbine 25 mg/m^2/day, days 1 and 8 every 21 days X 3
  Other Names: navelbine
  Arms: cisplatin/vinorelbine/docetaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Randomized phase II trial to study the effectiveness of two different combination chemotherapy regimens in treating patients who have stage IIIB or stage IV non-small cell lung cancer

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the survival and failure free survival of patients with advanced primary non-small cell lung cancer treated with carboplatin and gemcitabine followed by paclitaxel OR cisplatin and vinorelbine followed by docetaxel. II. Evaluate the response (confirmed plus unconfirmed) and toxicities associated with these two regimens in these patients.

OUTLINE: This is a randomized study. Patients are randomized to one of two treatment arms. Arm I: Patients receive carboplatin IV over 30 minutes on day 1 followed by gemcitabine IV over 30 minutes on days 1 and 8. Treatment repeats every 21 days for 3 courses. Following the 3 courses of carboplatin and gemcitabine, patients receive paclitaxel IV over 3 hours on day 1 every 21 days for 3 courses. Arm II: Patients receive cisplatin IV over 30-60 minutes on day 1 followed by vinorelbine IV over 6-10 minutes on days 1 and 8. Treatment repeats every 21 days for 3 courses. Following the 3 courses of cisplatin and vinorelbine, patients receive docetaxel IV over 1 hour on day 1 every 21 days for 3 courses. Patients receive no further treatment until evidence of disease progression. Patients are followed every 2 months for the first year, every 6 months for years 2 and 3, and annually thereafter.

PROJECTED ACCRUAL: A total of 160 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed newly diagnosed stage IIIB or IV advanced primary non-small cell lung cancer (adenocarcinoma, large cell carcinoma, squamous cell carcinoma, or unspecified) or recurrent non-small cell lung cancer after previous surgery and/or radiotherapy Stage IIIB: T4 lesion due to malignant pleural effusion, OR multiple lesions in a single lobe containing a T3 or T4 primary, OR lesions in multiple lobes of the ipsilateral lung for which one such lesion is T3 or T4 Any N M0 Stage IV: Any T, Any N, M1 Measurable or evaluable disease Measurable or evaluable disease must be outside of the prior radiotherapy port or prior surgical resection area No brain metastases No bronchoalveolar carcinoma or stage IIIB tumor involving the superior sulcus (pancoast tumors)

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: SWOG 0-1 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Creatinine no greater than 2 times upper limit of normal AND Creatinine clearance at least 50 mL/min Other: No prior malignancy in the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or adequately treated stage I or II cancer from which the patient is currently in complete remission Not pregnant or nursing Effective contraception required of all fertile patients

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior biologic therapy for non-small cell lung cancer No concurrent biologic therapy to measurable or evaluable lesions Chemotherapy: No prior systemic chemotherapy for non-small cell lung cancer Endocrine therapy: No concurrent hormonal therapy to measurable or evaluable lesions Radiotherapy: At least 3 weeks since prior radiotherapy and recovered No concurrent radiotherapy to measurable lesions Palliative radiation to small field nonmeasurable sites of disease (painful bony metastases) allowed Surgery: At least 3 weeks since surgery (thoracic or other major surgeries) and recovered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 1998-10; Primary Completion 2001-01 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin J. Edelman, MD, Study Chair — Veterans Affairs Medical Center - Baltimore
Locations (84):
- United States (84):
  - MBCCOP - University of South Alabama, Mobile, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock (McClellan), Little Rock, Arkansas
  - Beckman Research Institute, City of Hope, Duarte, California
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - University of California Davis Medical Center, Sacramento, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - University of Colorado Cancer Center, Denver, Colorado
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Dwight David Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Veterans Affairs Medical Center - Hines (Hines Junior VA Hospital), Hines, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - CCOP - Central Illinois, Springfield, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - MBCCOP - LSU Medical Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Veterans Affairs Medical Center - New Orleans, New Orleans, Louisiana
  - Louisiana State University Hospital - Shreveport, Shreveport, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - CCOP - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Providence Hospital - Southfield, Southfield, Michigan
  - Veterans Affairs Medical Center - Biloxi, Biloxi, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Ozarks Regional, Springfield, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - University of New Mexico Cancer Research & Treatment Center, Albuquerque, New Mexico
  - Veterans Affairs Medical Center - Brooklyn, Brooklyn, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Oklahoma City, Oklahoma City, Oklahoma
  - Oregon Cancer Center at Oregon Health Sciences University, Portland, Oregon
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - CCOP - Columbia River Program, Portland, Oregon
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Texas Tech University Health Science Center, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Swedish Hospital Tumor Institute, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington

REFERENCES:
- [Background] Lara PN Jr, Redman MW, Kelly K, Edelman MJ, Williamson SK, Crowley JJ, Gandara DR; Southwest Oncology Group. Disease control rate at 8 weeks predicts clinical benefit in advanced non-small-cell lung cancer: results from Southwest Oncology Group randomized trials. J Clin Oncol. 2008 Jan 20;26(3):463-7. doi: 10.1200/JCO.2007.13.0344. PMID 18202421
- [Background] Lara PN Jr, Redman MW, Kelly K, et al.: Alternative measures predicting clinical benefit in advanced non-small cell lung cancer (NSCLC) from Southwest Oncology Group (SWOG) randomized trials: implications for clinical trial design. [Abstract] J Clin Oncol 24 (Suppl 18): A-7006, 365s, 2006.
- [Result] Edelman MJ, Clark JI, Chansky K, Albain K, Bhoopalam N, Weiss GR, Giguere JK, Kelly K, Crowley J, Gandara DR. Randomized phase II trial of sequential chemotherapy in advanced non-small cell lung cancer (SWOG 9806): carboplatin/gemcitabine followed by paclitaxel or cisplatin/vinorelbine followed by docetaxel. Clin Cancer Res. 2004 Aug 1;10(15):5022-6. doi: 10.1158/1078-0432.CCR-04-0002. PMID 15297403
- [Result] Edelman MJ, Clark JI, Chansky K, et al.: Randomized phase II trial of sequential chemotherpy in advanced non-small cell lung cancer (SWOG 9806): carboplatin/gemcitabine (CARB/G) followed by paclitaxel (P) or cisplatin/vinorelbine (C/V) followed by docetaxel (D). [Abstract] Proceedings of the American Society of Clinical Oncology 20: A-1254, 314, 2001.